CLINICAL TRIAL: NCT03994601
Title: A Phase 1/2 First-in-human Study of BMS-986288 Alone and in Combination With Nivolumab in Advanced Malignant Tumors
Brief Title: An Investigational Immunotherapy Study of BMS-986288 Alone and in Combination With Nivolumab in Advanced Solid Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA043-001; 2021-004284-27 (EudraCT Number)
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: BMS-986288 Monotherapy (Experimental)
  Interventions: Drug: BMS-986288
- Arm B: BMS-986288 in combination with Nivolumab (Experimental)
  Interventions: Drug: BMS-986288; Drug: Nivolumab
- Part 2C: BMS-986288 in combination with Nivolumab and Regorafenib (Experimental)
  Interventions: Drug: BMS-986288; Drug: Nivolumab; Drug: Regorafenib

INTERVENTIONS:
Drug: BMS-986288 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm B: BMS-986288 in combination with Nivolumab; Part 2C: BMS-986288 in combination with Nivolumab and Regorafenib
Drug: Regorafenib — Specified dose on specified days
  Arms: Part 2C: BMS-986288 in combination with Nivolumab and Regorafenib

SUMMARY:
The purpose of this study is to determine whether BMS-986288 both by itself and in combination with Nivolumab is safe and tolerable in the treatment of select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of select solid tumor that is advanced (metastatic, recurrent, and/or unresectable) with measurable disease and have at least 1 lesion accessible for biopsy
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Received, and then progressed, relapsed, or been intolerant to, at least 1 standard treatment regimen in the advanced or metastatic setting according to select solid tumor histologies

Exclusion Criteria:

* Active, known or suspected autoimmune disease
* Active malignancy requiring concurrent intervention
* Primary Central Nervous System (CNS) malignancies or tumors with CNS metastasis as the only site of disease, will be excluded

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- United States (6):
  - Local Institution - 0075, Costa Mesa, California
  - Local Institution - 0050, Orange, California
  - Local Institution - 0005, Aurora, Colorado
  - Local Institution - 0002, Baltimore, Maryland
  - Local Institution - 0004, St Louis, Missouri
  - Local Institution - 0001, Hackensack, New Jersey
- Argentina (8):
  - Local Institution - 0011, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0074, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0014, Córdoba, Córdoba Province
  - Local Institution - 0013, Río Cuarto, Córdoba Province
  - Local Institution - 0008, ABB, Distrito Federal
  - Local Institution - 0012, CABA, Distrito Federal
  - Local Institution - 0017, Buenos Aires
  - Local Institution - 0016, Buenos Aires
- Canada (3):
  - Local Institution - 0006, Toronto, Ontario
  - Local Institution - 0042, Montreal, Quebec
  - Local Institution - 0046, Montreal, Quebec
- Chile (5):
  - Local Institution - 0010, Viña del Mar, Región de Valparaíso
  - Local Institution - 0036, Santiago, Santiago Metropolitan
  - Local Institution - 0019, Santiago, Santiago Metropolitan
  - Local Institution - 0035, Santiago, Santiago Metropolitan
  - Local Institution - 0009, Santiago, Santiago Metropolitan
- France (6):
  - Local Institution - 0034, Bordeaux, Gironde
  - Local Institution - 0022, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0018, Bron
  - Local Institution - 0026, Marseille
  - Local Institution - 0015, Paris
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon
- Italy (6):
  - Local Institution - 0040, Milan, Lombardy
  - Local Institution - 0038, Padua, Veneto
  - Local Institution - 0028, Ancona
  - Local Institution - 0033, Catanzaro
  - Local Institution - 0031, Milan
  - Local Institution - 0039, Roma
- Spain (6):
  - Local Institution - 0056, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0054, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0023, Madrid
  - Local Institution - 0024, Majadahonda
  - Local Institution - 0055, Seville
  - Local Institution - 0025, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1A: Cohort 1: BMS-986288 BMS 20mg Q4W
- Treatment 1A: Cohort 2: BMS-986288 40mg Q4W
- Treatment 1A: Cohort 3: BMS-986288 80mg Q4W
- Treatment 1A: Cohort 4: BMS-986288 160mg Q4W
- Treatment 1A: Cohort 5: BMS-986288 320mg Q4W
- Treatment 1A: Cohort 6: BMS-986288 480mg Q4W
- Treatment 1B: Cohort 1; Treatment 2B: Cohort 1: BMS-986288 80mg + Nivo 480mg Q4W
- Treatment 1B: Cohort 2; Treatment 2B: Cohort 2; Treatment 2C: Cohort 1: BMS-986288 120mg + Nivo 480mg Q4W
- Treatment 1B: Cohort 3: BMS-986288 160mg + Nivo 480mg Q4W
- Treatment 2C: Cohort 2: Regorafenib 160mg PO QD first 21 days of 28-day cycle
Period: Overall Study
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2 | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2
Started | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39 | 34 | 12
Crossing Over (Crossing over to Treatment 2C: Cohort 3 (BMS-986288 120mg + Nivo 480mg Q4W)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Option to crossing over to Treatment 2C: Cohort 3 due to disease progression)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39 | 33 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 7 | 4 | 1 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 4 | 1 | 3
Not completed — Other Reasons | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 4 | 3 | 4 | 2
Not completed — Disease Progression | 3 | 3 | 4 | 6 | 3 | 5 | 7 | 25 | 1 | 24 | 20 | 24 | 7
Not completed — Study Drug Toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 3 | 0
Not completed — AE Unrelated to Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 5 | 0 | 0
Not completed — Request to Discontinue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2 | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Total
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39 | 34 | 12 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (18.10) | 61.3 (7.46) | 63.4 (9.37) | 65.3 (8.71) | 58.8 (5.40) | 54.8 (13.59) | 66.2 (10.76) | 59.6 (11.63) | 69.7 (6.66) | 63.3 (9.44) | 64.7 (8.09) | 61.2 (11.43) | 59.4 (8.45) | 61.9 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 2 | 4 | 17 | 2 | 14 | 11 | 14 | 5 | 79
  Male | 2 | 1 | 3 | 5 | 3 | 3 | 5 | 23 | 1 | 33 | 28 | 20 | 7 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 6 | 4 | 9 | 3 | 28
  Not Hispanic or Latino | 3 | 4 | 4 | 5 | 4 | 5 | 7 | 28 | 1 | 8 | 17 | 10 | 4 | 100
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 9 | 1 | 33 | 18 | 15 | 5 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 7
  White | 3 | 1 | 3 | 5 | 5 | 5 | 8 | 33 | 2 | 44 | 38 | 33 | 11 | 191
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety Related Events for Cohorts 1A, 1B and 2B.
Description: Safety releated events for Cohorts 1A, 1B and 2B.
Time Frame: approximately 6 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39
Participants
  AEs | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39
  SAEs | 3 | 3 | 4 | 3 | 5 | 5 | 4 | 29 | 3 | 34 | 30
  AEs Leading to Discontinuation | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 12 | 2 | 14 | 15
  Deaths | 3 | 4 | 5 | 2 | 3 | 5 | 5 | 26 | 2 | 34 | 30

2. Primary Outcome: Dose Limiting Toxicities Cohorts 1A, 1B and 2B.
Description: A DLT is an adverse event or abnormal lab value not related to disease progression, illness, or other medications. The DLT evaluation period is 5 weeks (35 days) for both BMS-986288 monotherapy and combination dose escalation. Toxicities beyond this period will inform final dose decisions. Participants who discontinue due to a DLT or complete the 5-week period after receiving at least 2 doses are considered DLT-evaluable. Those who withdraw early or receive fewer than 2 doses for non-DLT reasons are not evaluable and may be replaced. Participants with dose delays for non-DLT reasons remain evaluable if they receive at least 2 doses within 8 weeks.
Time Frame: approximately 5 weeks
Population: As Per Protocol, DLT Evaluable Participants in 1A, 1B and 2B.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 4 | 2 | 6 | 19 | 3 | 0 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2

3. Primary Outcome: Objective Response Rate by BICR in Cohort 2C
Description: The percentage of all treated participants whose BOR is either CR or PR by BICR per RECIST v1.1.
Time Frame: approximately 2.15 Months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage or Participants
Groups:
- Treatment 2C: Cohort 3: BMS-986288 120mg + Nivo 480mg Q4W (Crossover from Treatment 2C: Cohort 2)
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Percentage or Participants | 0 [0.0 to 10.3] | 0 [0.0 to 26.5] | 0 [0.0 to 60.2]

4. Secondary Outcome: Objective Response Rate in Cohorts 1A, 1B and 2B
Description: The percentage of all treated participants whose BOR is either CR or PR by Investigator per RECIST v1.1.
Time Frame: approximately 2.15 Months
Population: All Treated Participants in Cohort 1A, 1B and 2B
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39
Percentage of Participants | 0 [0.0 to 60.2] | 25.0 [0.6 to 80.6] | 20.0 [0.5 to 71.6] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2] | 22.2 [2.8 to 60.0] | 5.0 [0.6 to 16.9] | 0 [0.0 to 70.8] | 6.4 [1.3 to 17.5] | 7.7 [1.6 to 20.9]

5. Secondary Outcome: Duration of Response in Cohorts 1A, 1B and 2B
Description: Duration of response is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the 1st objectively documented tumor progression as determined by Investigator (per RECIST 1.1), or death due to any cause, whichever occurs first.
Time Frame: approximately 2.15 Months
Population: All Treated Participants in Cohort 1A, 1B and 2B who achievied CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 3
months |  | 5.68 [NA to NA] — insufficient number of participants with events to calculate via KM methodology | 5.59 [NA to NA] — insufficient number of participants with events to calculate via KM methodology |  |  |  | NA [3.12 to NA] — insufficient number of participants with events to calculate via KM methodology | NA [NA to NA] — insufficient number of participants with events to calculate via KM methodology |  | NA [2.73 to NA] — insufficient number of participants with events to calculate via KM methodology | 7.16 [5.91 to NA] — insufficient number of participants with events to calculate via KM methodology

6. Secondary Outcome: Time to Response in Cohorts 1A, 1B and 2B
Description: Time to response (TTR) assessed by investigator is defined as the time between the date of randomization and the first confirmed documented response (CR or PR) per RECIST 1.1 criteria.
Time Frame: approximately 2.15 Months
Population: All Treated Participants in Cohort 1A, 1B and 2B who achievied CR or PR
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 3
months |  | 1.64 (NA) — insufficient number of participants to calculate SD | 1.87 (NA) — insufficient number of participants to calculate SD |  |  |  | 4.78 (2.21) | 2.56 (1.30) |  | 6.14 (2.19) | 3.76 (3.45)

7. Secondary Outcome: Progression Free Survival in Cohorts 1A, 1B and 2B
Description: PFS is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression by investigator or death due to any cause, whichever is earlier.
Time Frame: approximately 2.15 Months
Population: All Treated Participants in Cohort 1A, 1B and 2B
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 6 | 5 | 5 | 9 | 40 | 3 | 47 | 39
Months | 1.05 [0.95 to NA] — insufficient number of participants with events to calculate via KM methodology | 1.49 [1.25 to NA] — insufficient number of participants with events to calculate via KM methodology | 1.68 [0.92 to NA] — insufficient number of participants with events to calculate via KM methodology | 4.65 [0.49 to NA] — insufficient number of participants with events to calculate via KM methodology | 1.81 [1.18 to NA] — insufficient number of participants with events to calculate via KM methodology | 1.15 [0.56 to NA] — insufficient number of participants with events to calculate via KM methodology | 1.76 [0.79 to 9.43] | 1.91 [1.75 to 2.46] | 1.71 [1.28 to NA] — insufficient number of participants with events to calculate via KM methodology | 2.63 [1.87 to 3.71] | 2.40 [1.91 to 3.78]

8. Secondary Outcome: Duration of Response by BICR in Cohort 2C
Description: Duration of response is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the 1st objectively documented tumor progression as determined by BICR (per RECIST 1.1), or death due to any cause, whichever occurs first.
Time Frame: approximately 2.5 Months
Population: All Treated Participants in Cohort 2C who achievied CR or PR
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: PFS by BICR in Cohort 2C
Description: PFS is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression by BICR or death due to any cause, whichever is earlier.
Time Frame: approximately 2.5 Months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Months | 2.10 [1.94 to 3.12] | 4.37 [1.74 to NA] — insufficient number of participants with events to calculate via KM methodology | 2.89 [1.87 to NA] — insufficient number of participants with events to calculate via KM methodology

10. Secondary Outcome: Overall Survival in Cohort 2C
Description: OS is defined as the time from randomization to the time of death due to any cause.
Time Frame: approximately 2.5 Months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Months | NA [4.67 to NA] — insufficient number of participants with events to calculate via KM methodology | 6.67 [4.37 to NA] — insufficient number of participants with events to calculate via KM methodology | NA [6.37 to NA] — insufficient number of participants with events to calculate via KM methodology

11. Secondary Outcome: Objective Response Rate by Investigator in Cohort 2C
Description: The percentage of all treated participants whose BOR is either CR or PR by Investigator per RECIST v1.1.
Time Frame: approximately 2.5 Months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage or Participants
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Percentage or Participants | 0 [0.0 to 10.3] | 0 [0.0 to 26.5] | 0 [0.0 to 60.2]

12. Secondary Outcome: Duration of Response by Investigator in Cohort 2C
Description: as for outcome 5
Time Frame: approximately 2.5 Months
Population: All Treated Participants in Cohort 2C who achievied CR or PR
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: PFS by Investigator in Cohort 2C
Description: as for outcome 7
Time Frame: approximately 2.5 Months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Months | 2.04 [1.91 to 2.40] | 4.37 [1.91 to 5.32] | 2.89 [1.87 to NA] — insufficient number of participants with events to calculate via KM methodology

14. Secondary Outcome: Safety Related Events in Cohort 2C
Description: Safety Related Events in Cohort 2C
Time Frame: approximately 6 Months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 34 | 12 | 4
Participants
  AEs | 34 | 12 | 4
  SAEs | 24 | 7 | 3
  AEs leading to discontinuation | 5 | 2 | 0
  Deaths | 12 | 6 | 1

15. Secondary Outcome: Dose Limiting Toxicities in Cohort 2C
Description: as for outcome 2
Time Frame: approximately 5 weeks
Population: As Per Protocol, DLT Evaluable Participants in 2C.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
Number analyzed (Participants) | 8 | 1 | 1
Participants | 0 | 0 | 0

16. Secondary Outcome: Cmax for Cohorts 1A, 1B and 2B
Description: Cmax is defined as maximum plasma concentration of the drug.
Time Frame: On Cycle 1 Day 1 for Total and Intact, C4D1 for Intact
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 5 | 5 | 9 | 40 | 3 | 44 | 37
ng/mL
  Total; C1D1 | 7346.016 (121.526) | 10146.620 (54.040) | 23583.104 (15.499) | 35151.545 (18.956) | 80443.781 (19.688) | 118980.802 (12.916) | 18536.692 (29.410) | 32373.657 (27.926) | 49789.464 (16.011) | 24029.527 (29.190) | 33140.927 (30.622)
  Intact; C1D1 | 7308.897 (116.031) | 9260.703 (50.656) | 23165.692 (13.694) | 37136.774 (18.071) | 80597.586 (20.770) | 116519.624 (18.629) | 19623.300 (30.309) | 33312.894 (25.718) | 43461.861 (19.858) | 24507.324 (29.670) | 34865.711 (32.039)
  Intact, C4D1: number analyzed (Participants) | 0 | 1 | 2 | 4 | 0 | 0 | 3 | 12 | 0 | 19 | 10
  Intact, C4D1 |  | 16700.000 (NA) — Insufficient number of participants for calculation of %GeoCV | 25674.890 (31.915) | 32697.980 (27.325) |  |  | 24303.414 (20.997) | 30897.984 (19.853) |  | 24900.543 (30.863) | 29962.683 (39.665)

17. Secondary Outcome: Tmax for Cohorts 1A, 1B and 2B
Description: Tmax is defined is the time to maximum plasma concentration
Time Frame: On Cycle 1 Day 1 for Total and Intact, C4D1 for Intact
Population: PK Evaluable Population
Measure: Median (Full Range); unit: Hours (H)
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 5 | 5 | 9 | 40 | 3 | 44 | 37
Hours (H)
  Total; C1D1 | 2.500 [0.52 to 76.25] | 3.725 [0.62 to 21.50] | 0.833 [0.62 to 4.50] | 4.00 [0.97 to 4.50] | 4.00 [1.00 to 24.47] | 3.983 [1.00 to 4.00] | 2.933 [0.50 to 3.07] | 2.758 [0.52 to 23.72] | 3.000 [2.87 to 4.50] | 1.100 [0.50 to 69.08] | 2.800 [0.62 to 163.83]
  Intact; C1D1 | 2.500 [0.52 to 76.25] | 3.725 [0.62 to 4.75] | 4.100 [0.50 to 4.60] | 4.000 [0.70 to 4.50] | 1.000 [0.97 to 5.02] | 4.000 [1.00 to 4.00] | 2.933 [0.50 to 3.07] | 2.584 [0.52 to 23.72] | 0.567 [0.53 to 4.50] | 1.109 [0.52 to 69.08] | 2.683 [0.50 to 67.25]
  Intact; C4D1: number analyzed (Participants) | 0 | 1 | 2 | 4 | 0 | 0 | 3 | 12 | 0 | 19 | 10
  Intact; C4D1 |  | 0.80 [0.80 to 0.80] | 2.609 [0.60 to 4.62] | 4.000 [4.00 to 4.03] |  |  | 2.917 [0.57 to 2.92] | 1.175 [0.50 to 3.00] |  | 1.067 [0.10 to 22.27] | 1.942 [0.50 to 163.92]

18. Secondary Outcome: AUC(0-T) for Cohorts 1A, 1B and 2B
Description: Area under the plasma concentration time-curve. AUC from time 0 to the last time of quantifiable concentration.
Time Frame: On Cycle 1 Day 1 for Total and Intact, C4D1 for Intact
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*ng/mL
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 5 | 5 | 9 | 40 | 3 | 44 | 37
H*ng/mL
  Total; C1D1 | 1082346.14014 (75.57449) | 1861226.97707 (64.94566) | 4508154.21783 (26.12088) | 6723961.51187 (34.12795) | 15142162.8434 (16.00843) | 22403650.45029 (1.36445) | 3703077.82498 (42.06667) | 5353398.24303 (37.21041) | 10304729.49651 (12.43122) | 4076700.36940 (37.12350) | 5722320.50118 (33.73607)
  Intact C1D1 | 896640.17927 (69.08315) | 1351357.71064 (50.85821) | 3347814.86599 (24.70946) | 5142468.12364 (32.63080) | 10800750.41369 (24.56514) | 16484408.30096 (32.66786) | 2741905.79748 (44.37964) | 4235280.11485 (35.64573) | 6885601.91062 (16.07058) | 3132449.17983 (36.23668) | 4572710.36078 (31.51764)
  Intact C4D1: number analyzed (Participants) | 0 | 1 | 2 | 4 | 0 | 0 | 3 | 12 | 0 | 19 | 10
  Intact C4D1 |  | 2497426.80175 (NA) — Insufficient number of events to calculate %GeoCV | 4054657.85996 (32.35490) | 3130520.59300 (174.06709) |  |  | 4426043.81234 (29.52488) | 3519951.91889 (82.74941) |  | 2693455.25993 (160.22857) | 4971148.07876 (36.10988)

19. Secondary Outcome: AUC(Tau) for Cohorts 1A, 1B and 2B
Description: Area under the plasma concentration time-curve. AUC over the dosing interval.
Time Frame: On Cycle 1 Day 1 for Total and Intact, C4D1 for Intact
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*ng/mL
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 5 | 5 | 9 | 39 | 3 | 44 | 35
H*ng/mL
  Total; C1D1 | 1331755.67815 (60.64583) | 2264731.07676 (42.75268) | 4605903.87150 (24.90666) | 6723961.51187 (34.12795) | 16182654.45947 (11.93735) | 23790801.57085 (2544267) | 3918392.93186 (36.00362) | 5591689.93928 (31.50690) | 10304729.49651 (12.43122) | 4322664.92642 (30.29295) | 5910861.95661 (31.50360)
  Intact; C1D1 | 1010308.46356 (56.80904) | 1442135.68976 (46.75056) | 3385414.54789 (24.62737) | 5142468.12364 (32.63080) | 11352433.48069 (22.51990) | 17091968.12404 (30.59115) | 289264.80314 (40.11934) | 4377298.23824 (31.63194) | 6885601.91062 (16.07058) | 3293311.90482 (31.99041) | 4712874.56281 (31.65019)
  Intact; C4D1: number analyzed (Participants) | 0 | 1 | 2 | 3 | 0 | 0 | 3 | 11 | 0 | 18 | 10
  Intact; C4D1 |  | 2497426.80175 (NA) — Insufficient number of events to calculate %GeoCV | 4163018.66565 (28.37040) | 6019278.27350 (16.21812) |  |  | 4426043.81234 (29.52488) | 4400418.11940 (29.49927) |  | 3520845.93694 (26.05394) | 5016568.84128 (33.17484)

20. Secondary Outcome: C(Tau) for Cohorts 1A, 1B and 2B
Description: Ctau is defined as the concentration of study drug at the end of the dosing interval
Time Frame: On Cycle 1 Day 1 for Total and Intact, C4D1 for Intact
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 4 | 9 | 40 | 3 | 47 | 39
ng/mL
  Total; C1D1 | 323.28443 (235.05609) | 1255.33355 (55.24318) | 2756.28704 (51.54927) | 3459.203 (53.635) | 7295.79216 (30.41409) | 12665.79193 (35.88453) | 1968.67090 (86.25269) | 2006.56628 (79.18517) | 5541.408 (29.721) | 1855.23484 (91.20240) | 2204.14352 (66.31300)
  Intact: C1D1: number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 4 | 9 | 39 | 3 | 43 | 32
  Intact: C1D1 | 131.78635 (184.60547) | 364.39683 (100.05639) | 1024.74019 (78.02372) | 1423.007 (72.743) | 2496.26953 (57.42368) | 4683.23900 (44.94995) | 732.11636 (119.96752) | 765.14910 (112.89925) | 5145.910 (22.999) | 799.46828 (95.65148) | 935.75687 (91.60647)
  Intact; C4D1: number analyzed (Participants) | 0 | 1 | 2 | 3 | 0 | 0 | 3 | 9 | 0 | 18 | 8
  Intact; C4D1 |  | 687.000 (NA) — Insufficient number of events to calculate %GeoCv | 1365.54472 (118.69550) | 2082.90863 (41.58557) |  |  | 1940.311 (33.795) | 1123.88313 (87368335) |  | 907.65893 (76.11507) | 1155.32105 (64.19719)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: Approximately 6 Months All-Cause mortality (From randomization to end of study): Approximately 5 years
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment 1A: Cohort 1 | Treatment 1A: Cohort 2 | Treatment 1A: Cohort 3 | Treatment 1A: Cohort 4 | Treatment 1A: Cohort 5 | Treatment 1A: Cohort 6 | Treatment 1B: Cohort 1 | Treatment 1B: Cohort 2 | Treatment 1B: Cohort 3 | Treatment 2B: Cohort 1 | Treatment 2B: Cohort 2 | Treatment 2C: Cohort 1 | Treatment 2C: Cohort 2 | Treatment 2C: Cohort 3
All-Cause Mortality (participants affected / at risk) | 3/4 | 4/4 | 5/5 | 2/6 | 3/5 | 5/5 | 5/9 | 26/40 | 2/3 | 34/47 | 30/39 | 12/34 | 6/12 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 4/5 | 3/6 | 5/5 | 5/5 | 4/9 | 29/40 | 3/3 | 34/47 | 30/39 | 24/34 | 7/12 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 6/6 | 5/5 | 5/5 | 9/9 | 40/40 | 3/3 | 47/47 | 39/39 | 34/34 | 12/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1A: Cohort 1 (N=4) | Treatment 1A: Cohort 2 (N=4) | Treatment 1A: Cohort 3 (N=5) | Treatment 1A: Cohort 4 (N=6) | Treatment 1A: Cohort 5 (N=5) | Treatment 1A: Cohort 6 (N=5) | Treatment 1B: Cohort 1 (N=9) | Treatment 1B: Cohort 2 (N=40) | Treatment 1B: Cohort 3 (N=3) | Treatment 2B: Cohort 1 (N=47) | Treatment 2B: Cohort 2 (N=39) | Treatment 2C: Cohort 1 (N=34) | Treatment 2C: Cohort 2 (N=12) | Treatment 2C: Cohort 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 4 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 4 | 4 | 1 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1 | 2 | 4 | 1 | 10 | 2 | 13 | 8 | 5 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 5 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Assisted suicide (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1A: Cohort 1 (N=4) | Treatment 1A: Cohort 2 (N=4) | Treatment 1A: Cohort 3 (N=5) | Treatment 1A: Cohort 4 (N=6) | Treatment 1A: Cohort 5 (N=5) | Treatment 1A: Cohort 6 (N=5) | Treatment 1B: Cohort 1 (N=9) | Treatment 1B: Cohort 2 (N=40) | Treatment 1B: Cohort 3 (N=3) | Treatment 2B: Cohort 1 (N=47) | Treatment 2B: Cohort 2 (N=39) | Treatment 2C: Cohort 1 (N=34) | Treatment 2C: Cohort 2 (N=12) | Treatment 2C: Cohort 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 15 | 1 | 11 | 6 | 17 | 6 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 3 | 2 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5 | 0 | 0 | 2 | 1 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 2 | 6 | 6 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 2 | 0 | 4 | 13 | 0 | 18 | 6 | 12 | 6 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 1 | 2 | 1 | 8 | 0 | 7 | 6 | 6 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 3 | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 5 | 4 | 4 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 12 | 9 | 4 | 4 | 2
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 2 | 3 | 1 | 4 | 10 | 0 | 12 | 9 | 11 | 6 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 3 | 1 | 3 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 9 | 6 | 7 | 4 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pilonidal disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 4 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 9 | 1 | 2 | 4 | 8 | 4 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 5 | 1 | 2 | 2 | 6 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 12 | 1 | 0 | 5 | 14 | 7 | 2
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 8 | 4 | 8 | 2 | 0
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 1 | 1 | 0
Blood bilirubin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 0 | 2 | 2 | 7 | 6 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 9 | 2 | 6 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 8 | 1 | 4 | 1 | 6 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 2 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 3 | 1 | 3 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 3 | 2 | 1 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 5 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Coagulation test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 1 | 1 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 9 | 1 | 5 | 5 | 8 | 3 | 2
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5 | 0 | 11 | 4 | 7 | 3 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 9 | 0 | 12 | 6 | 7 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 3 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 1 | 2 | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 4 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 9 | 0 | 5 | 1 | 2 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 5 | 5 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 4 | 3 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fine motor skill dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 7 | 3 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 4 | 3 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 3 | 7 | 1 | 8 | 4 | 7 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 6 | 0 | 5 | 5 | 4 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 3 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 6 | 3 | 4 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 3 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 2 | 2 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 3 | 4 | 7 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03994601/Prot_SAP_000.pdf